CLINICAL TRIAL: NCT06808204
Title: Quality of Life Before and After Transcatheter Ablation in Children With Arrythmias
Acronym: QUALICATRYTHM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL24_0830; 2024-A02568-39 (Other: ID-RCB)
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Arrhythmia
Keywords: children; arrythmia; transcatheter ablation; quality of life
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children from 5 t17 years old suffering for arrythmia who need a transcatheter ablation (Experimental)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Quality of life questionnaire : Peds QL 4.0 (Pediatric Quality of Life )
Other: questionnaire — Physical activity level : Ricci and Gagnon questionnaire
Other: questionnaire — Anxiety questionnaire : State and Trait Inventory
Other: questionnaire — Depression questionnaire : Child Depression Inventory
Other: questionnaire — Child Depression Inventory
Other: questionnaire — Quality of life of parents before and after transcatheter ablation

SUMMARY:
The goal of this clinical trial is to evaluate the improvement in the quality of life after the transcatheter ablation in children from 5 to 17 years old suffering for arrythmia who need a transcatheter ablation (according to PACES recommendations). The main question is:

• to evaluate an improvement in the quality of life in these children, according to different questionnaires?

Participants will answer some questionnaires to get a global evaluation of the quality of life:

* Peds QL 4.0
* Peds QL 4.0 by proxy, which will be completed by the parents
* Ricci and Gagnon questionnaire
* Child Depression Index
* State and Trait Anxiety Inventory

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8 to 17
* Patients with a rhythm disorder,
* Patients with indication for catheter ablation according to PACES (Pediatric and Congenital Electrophysiology Society) recommendations,
* Patients and/or their parents/legal guardians who have given their non-objection to the study.

Exclusion Criteria:

* Refusal of child or parents/legal guardians
* Unability to understand and/or fill the quality of life questionnaire

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life before and after transcatheter ablation | one day before transcatheter ablation
  Quality of life before and after transcatheter ablation according to Quality of Life Inventory paediatrics (PedsQL) version 4.0 questionnaire.
  The questionnaire consists of 23 questions covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is used for the young child self-report (ages 5 to 7) (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem).
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate a better assessment of health-related quality of life.
Quality of life before and after transcatheter ablation | 3 months after transcatheter ablation
  Quality of life before and after transcatheter ablation according to Quality of Life Inventory paediatrics (PedsQL) version 4.0 questionnaire.
  The questionnaire consists of 23 questions covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is used for the young child self-report (ages 5 to 7) (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem).
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate a better assessment of health-related quality of life.
Quality of life before and after transcatheter ablation | 6 months after transcatheter ablation
  Quality of life before and after transcatheter ablation according to Quality of Life Inventory paediatrics (PedsQL) version 4.0 questionnaire.
  The questionnaire consists of 23 questions covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is used for the young child self-report (ages 5 to 7) (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem).
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate a better assessment of health-related quality of life.

SECONDARY OUTCOMES:
comparing level of activity before and after transcatheter ablation | one day before transcatheter ablation
  Level of activity before and after transcatheter ablation according to to the Ricci and Gagnon questionnaire.
  The self-assessment questionnaire is used to determine the patient's activity profile: inactive, active or very active. It consists of 9 questions with 5 suggested answers (giving a score from 1 to 5 for each answer given).
  The higher the score, the more active the profile (Less than 18 points in total: Inactive, Between 18 and 35 points in total: Active, More than 35 points in total: Very active).
comparing level of activity before and after transcatheter ablation | 3 months after transcatheter ablation
  Level of activity before and after transcatheter ablation according to to the Ricci and Gagnon questionnaire The self-assessment questionnaire is used to determine the patient's activity profile: inactive, active or very active. It consists of 9 questions with 5 suggested answers (giving a score from 1 to 5 for each answer given).
  The higher the score, the more active the profile (Less than 18 points in total: Inactive, Between 18 and 35 points in total: Active, More than 35 points in total: Very active).
comparing level of activity before and after transcatheter ablation | 6 months after transcatheter ablation
  Level of activity before and after transcatheter ablation according to to the Ricci and Gagnon questionnaire The self-assessment questionnaire is used to determine the patient's activity profile: inactive, active or very active. It consists of 9 questions with 5 suggested answers (giving a score from 1 to 5 for each answer given).
  The higher the score, the more active the profile (Less than 18 points in total: Inactive, Between 18 and 35 points in total: Active, More than 35 points in total: Very active).
comparing level of anxiety before and after transcatheter ablation | one day before transcatheter ablation
  Level of anxiety before and after transcatheter ablation according to the State-Trait Anxiety Inventory for Children (STAIC) questionnaire.
  The STAIC comprises 2 series of 20 items each: one concerns anxiety as a 'personality trait'; the other series concerns the subject's 'state of anxiety' at the time of completing the questionnaire, which may fluctuate over time.
  Each item is rated on a scale of 1 to 3. The overall score is obtained by a simple sum. The overall score varies between 20 and 60. The threshold score defining pathological anxiety is 34. The higher the score, the more anxious the patient.
comparing level of anxiety before and after transcatheter ablation | 3 months after transcatheter ablation
  Level of anxiety before and after transcatheter ablation according to the State-Trait Anxiety Inventory for Children (STAIC) questionnaire.
  The STAIC comprises 2 series of 20 items each: one concerns anxiety as a 'personality trait'; the other series concerns the subject's 'state of anxiety' at the time of completing the questionnaire, which may fluctuate over time.
  Each item is rated on a scale of 1 to 3. The overall score is obtained by a simple sum. The overall score varies between 20 and 60. The threshold score defining pathological anxiety is 34. The higher the score, the more anxious the patient.
comparing level of anxiety before and after transcatheter ablation | 6 months after transcatheter ablation
  Level of anxiety before and after transcatheter ablation according to the State-Trait Anxiety Inventory for Children (STAIC) questionnaire.
  The STAIC comprises 2 series of 20 items each: one concerns anxiety as a 'personality trait'; the other series concerns the subject's 'state of anxiety' at the time of completing the questionnaire, which may fluctuate over time.
  Each item is rated on a scale of 1 to 3. The overall score is obtained by a simple sum. The overall score varies between 20 and 60. The threshold score defining pathological anxiety is 34. The higher the score, the more anxious the patient.
comparing level of depression before and after transcatheter ablation | one day before transcatheter ablation
  Level of depression before and after transcatheter ablation according to the Child Depression Inventory (CDI) questionnaire.
  This questionnaire measures the intensity of depression in children and adolescents aged 7 to 17.
  Each item is scored from 0 (normal behaviour for age or absent) to 2 (severe). Adding the items together gives a total score of between 0 and 54. The higher the score, the more pathological the condition.
comparing level of depression before and after transcatheter ablation | 3 months after transcatheter ablation
  Level of depression before and after transcatheter ablation according to the Child Depression Inventory (CDI) questionnaire.
  This questionnaire measures the intensity of depression in children and adolescents aged 7 to 17.
  Each item is scored from 0 (normal behaviour for age or absent) to 2 (severe). Adding the items together gives a total score of between 0 and 54. The higher the score, the more pathological the condition.
comparing level of depression before and after transcatheter ablation | 6 months after transcatheter ablation
  Level of depression before and after transcatheter ablation according to the Child Depression Inventory (CDI) questionnaire.
  This questionnaire measures the intensity of depression in children and adolescents aged 7 to 17.
  Each item is scored from 0 (normal behaviour for age or absent) to 2 (severe). Adding the items together gives a total score of between 0 and 54. The higher the score, the more pathological the condition.
Quality of life of parents before and after transcatheter ablation | one day before transcatheter ablation
  Quality of life before and after transcatheter ablation according to PedsQL version 4.0 parents-kid questionnaire
  The questionnaire consists of 23 questions covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is used for the young child self-report (ages 5 to 7) (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem).
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate a better assessment of health-related quality of life.
Quality of life of parents before and after transcatheter ablation | 3 months after transcatheter ablation
  Quality of life before and after transcatheter ablation according to PedsQL version 4.0 parents-kid questionnaire
  The questionnaire consists of 23 questions covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is used for the young child self-report (ages 5 to 7) (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem).
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate a better assessment of health-related quality of life.
Quality of life of parents before and after transcatheter ablation | 6 months after transcatheter ablation
  Quality of life before and after transcatheter ablation according to PedsQL version 4.0 parents-kid questionnaire
  The questionnaire consists of 23 questions covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is used for the young child self-report (ages 5 to 7) (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem).
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3= 25, 4 = 0), so that higher scores indicate a better assessment of health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Francis BESSIERE, Dr, Principal Investigator — Hôpital cardiologique Louis Pradel - Hospices Civils de Lyon Service Rythmologie
Locations (7):
- France (7):
  - Hôpital cardiologique Louis Pradel, Bron
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Hôpital de la Timone, Marseille
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Cardiologique du Haut Lévêque - Service de cardiologie-électrophysiologie et stimulation cardiaque, Pessac
  - Hôpital Cardiologique du Haut Lévêque - Service des maladies cardio-vasculaires congénitales, Pessac
  - Clinique Pasteur, Toulouse